CLINICAL TRIAL: NCT05791123
Title: Alveolar Ridge Augmentation Following Tooth Extraction Using Bovine Xenograft With Platelet Rich Fibrin Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Medhat Sameh Abdelaziz, Assistant Lecturer of Prosthodontics, Future University in Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC-FDBSU/05012023-03/ER
Record Dates: First submitted 2023-03-08; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Bone Regeneration
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a bone graft mixed with PRF & covered by PRF membrane in fresh extraction socket (Experimental)
  Interventions: Procedure: a bone graft mixed with PRF & covered by PRF membrane in fresh extraction socket

INTERVENTIONS:
Procedure: a bone graft mixed with PRF & covered by PRF membrane in fresh extraction socket — Extraction sockets were filled with minced PRF clots mixed with the bovine xenograft and covered by PRF membranes to seal the extraction sockets.

SUMMARY:
fourteen patients requiring extraction of one posterior tooth with lost buccal bone (>50%) confirmed preoperatively by Cone-beam computed tomography (CBCT) scans. Extraction sockets were filled with minced PRF clots mixed with the bovine xenograft and covered by PRF membranes to seal the extraction sockets. (CBCT) scans, performed before tooth extraction and after 6 months, were used to assess vertical and horizontal bone changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients required implant treatment after tooth extraction
* Age group ranged from 20-60 years old.
* Patients could undergo the treatment under local anesthesia.
* Loss of buccal bone (>50%) confirmed by preoperative cone beam computed tomography (CBCT).
* Presence of other socket walls; mesial, distal and lingual walls.
* Tooth needed to be extracted in upper or lower posterior regions

Exclusion Criteria:

* Uncontrolled diabetic diseases.
* Uncontrolled hypertension, or hepatic and renal disorders.
* Any systemic diseases associated with bone metabolism.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
the change in alveolar bone width and height in mm using CBCT scans. | 6 months
  Cone Beam Computed Tomography were taken for each patients before tooth extraction and after 6 months, which were used to assess alveolar ridge changes in width and length in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, Egypt

REFERENCES:
- [Derived] Elbanna RM, Abdelaziz MS, Alameldeen HE. Augmentation of single tooth extraction socket with deficient buccal walls using bovine xenograft with platelet-rich fibrin membrane. BMC Oral Health. 2023 Nov 17;23(1):874. doi: 10.1186/s12903-023-03554-2. PMID 37978487